CLINICAL TRIAL: NCT04887324
Title: Real-life Data of Constitutional Von Willebrand Disease in Western France: Treatment Outcomes With the Recombinant Von Willebrand Factor
Brief Title: Real-life Data of Constitutional Von Willebrand Disease in Western France
Acronym: HOPSCOTCH-II
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0188
Record Dates: First submitted 2021-04-15; First posted 2021-05-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Von Willebrand Diseases
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The objective of this observational study HOPSCOTcH-WILL II is to provide an accurate and detailed account of current Von Willebrand Disease (VWD) therapeutic management by collecting real-life data on hemorrhagic treated events in the 5 Western French Hemophilia Treatment Center.

The HOPSCOTCH-WILL II study aims to describe therapeutic management of patients with VWD, following the provision of a recombinant drug in France; It will also permit to carry out a budget impact analysis to quantify the economic significance of this new era.

ELIGIBILITY:
Inclusion Criteria:

* Constitutional Von Willebrand Disease patient, of any severity, with or without Von Willebrand Factors inhibitors
* Patient included in the research database BERHLINGO
* Patient treated or not by desmopressin or Von Willebrand Factor/FVIII/by-passing agents available on the French market (at baseline)
* Patient who agrees to participate in the HOPSCOTcH-Will II and followed in one of the 5 investigator centers

Exclusion Criteria:

- Patients under guardianship

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Constitutional Von Willebrand Disease patients
Sampling Method: Non-Probability Sample
Enrollment: 922 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Observational study, description of the global therapeutic modalities required for severe treated hemorrhagic events in constitutional Von Willebrand Disease patients of any severity | 4 years
  Data collection for evaluation of Clotting factors quantities used by collection of treatments for severe hemorrhagic events

CONTACTS AND LOCATIONS:
Overall Officials: Marc Trossaert, Principal Investigator — Nantes University Hospital
Locations (5):
- France (5):
  - CHU Angers, Angers
  - CHR de Brest, Brest
  - CH Le Mans, Le Mans
  - CHU de Nantes, Nantes
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided